CLINICAL TRIAL: NCT03376633
Title: The Promise of a School-Based, Trauma-Informed Cognitive Behavioral Therapy Intervention for Young Women in Chicago: A Randomized Evaluation
Brief Title: The Impact of a School-Based, Trauma-Informed CBT Intervention for Young Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Northwestern University (Other); Youth Guidance (Unknown); Chicago Public Schools (Other); U.S. Department of Justice (U.S. Federal Agency); Paul M. Angell Family Foundation (Unknown); Polk Bros. Foundation (Unknown); The Reva & David Logan Foundation (Unknown); DePaul University (Other); Laura and John Arnold Foundation (Other); MacArthur Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB17-0585
Record Dates: First submitted 2017-12-04; First posted 2017-12-18 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Anxiety; Anxiety Disorders; Behavioral Symptoms; Depression; Mental Disorders; Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic; Trauma and Stressor Related Disorders; Wounds and Injuries
Keywords: Randomized Controlled Trial; RCT; Chicago Public Schools; high school; trauma-informed counseling; group-based counseling; counseling; mentoring; Cognitive Behavioral Therapy; CBT; adolescents; females; trauma; stress; PTSD; anxiety; depression; graduation
MeSH Terms: conditions — Anxiety Disorders; Behavioral Symptoms; Depression; Mental Disorders; Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic; Trauma and Stressor Related Disorders; Wounds and Injuries

STUDY DESIGN:
Masking Description: Treatment individuals will be provided information about the trial and consented into the study as part of WOW program materials (note: program participation is not conditional on participation in the research). Control individuals will not be provided information about the study, but may be provided information if they inquire about programming. Due to the intervention type, it is not possible to mask the identity of treatment participants from the provider or from participants. However, the provider will not be informed of the identity of the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): These youth will not receive Working on Womanhood (WOW) services during academic years 2017-18 and 2018-19 [Cohort 1] or 2018-19 and 2019-20 [Cohort 2] or after, and will not have contact with WOW clinicians. Control youth will be able to receive all other services available through their school as they normally would, such as access to the school counselor and after school programs.
- WOW Group and Individual Counseling (Experimental): These youth will receive Working on Womanhood (WOW) services during academic years 2017-18 and 2018-19 [Cohort 1] or 2018-19 and 2019-20 [Cohort 2]. These young women will participate in weekly group therapy and skill-building sessions, led by master's level clinicians, and will also receive individual support and therapy from their clinicians as-needed.
  Interventions: Behavioral: Working on Womanhood (WOW)

INTERVENTIONS:
Behavioral: Working on Womanhood (WOW) — A trauma-informed group counseling and clinical mentoring intervention for young women
  Arms: WOW Group and Individual Counseling

SUMMARY:
The purpose of this study is:

1. To conduct a randomized controlled trial to evaluate the impact of Working on Womanhood (WOW), a school-based, trauma-informed counseling and clinical mentoring program for young women in Chicago, on PTSD, anxiety, depression. In addition, this study will examine the effect of WOW on other, secondary outcomes such as school discipline, GPA, high school graduation, and criminal justice involvement, risky behaviors, and other social-emotional learning outcomes.
2. To evaluate the cost-effectiveness of the WOW program.

DETAILED DESCRIPTION:
The University of Chicago Crime Lab and Education Lab are partnering with the City of Chicago, Chicago Public Schools, and Youth Guidance to implement a randomized controlled trial to test the efficacy of Youth Guidance's Working on Womanhood program across two cohorts: Cohort 1, receiving programming during academic years 2017-18 and 2018-19, and Cohort 2, receiving programming during academic years 2018-19 and 2019-20. For Cohort 1, incoming 9th, 10th, and 11th grade female students in 10 Chicago Public Schools high schools (as of Fall 2017) will be screened for eligibility and randomized to either a treatment group that will be offered to receive WOW services over two academic years, or to a control group that will not be offered to receive WOW services over two academic years. For cohort 2, only incoming 9th graders (as of Fall 2018) will be randomized, in the same manner. Control group students will still be eligible to receive other status quo school and community supports. Outcomes of interest will be measured using administrative data and a comprehensive student survey.

WOW is a trauma-informed, in-school group counseling and clinical mentoring program developed by non-profit Youth Guidance. Informed by CBT, WOW helps girls challenge unhelpful thoughts and build self-esteem and self-efficacy to make positive and healthy decisions. WOW aims to reduce depression, anxiety, and PTSD symptoms, and improve academic and behavioral outcomes. WOW delivers a 26-lesson curriculum via weekly small-group counseling sessions during the school day. The curriculum is designed around five core values: self-awareness, emotional intelligence, healthy relationships, visionary goal setting, and leadership, and delivered by masters-level social workers and counselors. WOW counselors may also provide individual counseling and referrals to other services. The WOW program fills a critical gap in the existing set of programs available to these students, by providing services that cater to the unique needs of young women in our most under-resourced high schools.

ELIGIBILITY:
Inclusion Criteria:

* Chicago Public Schools high schools, chosen in collaboration with Youth Guidance leadership, that serve majority low-income, minority students in community areas impacted by violence
* School's 9th, 10th, and 11th grade female student population is large enough to support at least 50 treatment students and 50 control students, after accounting for a 60 to 70 percent take-up rate and exclusion criteria
* Schools do not currently have WOW services (as of AY2016-17)
* School administrators are enthusiastic about the program and agree to the terms and conditions of the experimental design
* All female students in these selected schools entering 9th, 10th, or 11th grade in Fall 2017, or entering 9th grade in Fall 2018.

Exclusion Criteria:

* Students with an overall attendance rate below 75% during AY2016-17 [Cohort 1] or AY2017-18 [Cohort 2]
* Students who display proactive aggression towards others
* Students with severe cognitive / developmental disabilities, these include: autistic, emotional and behavior disorder, educable mental handicap, intellectual disability - profound, severe/profound handicap, and trainable mental handicap

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 5106 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Change in depression assessment score | Up to 36 months
  Score on self-reported depression screen, obtained from the Behavior Assessment System for Children, Third Edition (BASC-3) Self-Report of Personality (SRP)
Change in post-traumatic stress disorder (PTSD) assessment score | Up to 36 months
  Score on self-reported PTSD screen, obtained from the Child and Adolescent Trauma Screen (CATS)
Change in anxiety assessment score | Up to 36 months
  Score on self-reported anxiety screen, obtained from the BASC-3 SRP

SECONDARY OUTCOMES:
Change in high school graduation | Up to 5 years
  On-time graduation rate, obtained from Chicago Public Schools (CPS) administrative database
Change in absences | 1-year, 2-year, 3-year, 4-year, 5-year
  Rate and number of school absences, obtained from CPS administrative database
Change in index of CPS schooling outcomes | 1-year, 2-year, 3-year, 4-year, 5-year
  Standardized index composed of GPA, number of course failures, attendance rate, and number of in-school and out-of-school suspensions, obtained from CPS administrative database
Change in student misconduct | 1-year, 2-year, 3-year, 4-year, 5-year
  Number of in-school and out-of-school suspensions, obtained from CPS administrative database
Change in course failures | 1-year, 2-year, 3-year, 4-year, 5-year
  Rate and number of courses failed, obtained from CPS administrative database
Change in overall arrests | 1-year, 2-year, 3-year, 4-year, 5-year
  Number of total arrests, obtained from Chicago Police Department (CPD) and Illinois State Police (ISP) administrative databases
Change in violent crime arrests | 1-year, 2-year, 3-year, 4-year, 5-year
  Number of arrests for violent crimes, obtained from CPD and ISP administrative databases
Change in other arrests (property, drug, and other) | 1-year, 2-year, 3-year, 4-year, 5-year
  Number of non-violent crime arrests, including property crimes, drug crimes, and other crimes, obtained from CPD and ISP administrative databases

OTHER OUTCOMES:
Change in pregnancy/childbirth rate | 1-year, 2-year, 3-year, 4-year, 5-year
  Self-reported survey measures, obtained from representative student survey; Childbirth data, obtained from the Chicago and Illinois Dept. of Public Health
Change in sexual health and behaviors | Up to 36 months
  Self-reported survey measures, obtained from representative student survey
Change in substance use | Up to 36 months
  Self-reported survey measures, obtained from representative student survey
Change in school attitudes and engagement | Up to 36 months
  Self-reported survey measures, obtained from representative student survey
Change in family cohesion | Up to 36 months
  Measures adapted from the Family Environment Scale (relationships section), obtained from representative student survey
Change in self-esteem (self-reliance, sense of inadequacy) | Up to 36 months
  Self-reported survey measures, obtained from representative student survey
Change in emotional regulation | Up to 36 months
  Score on the Difficulties in Emotion Regulation Scale - Short Form (DERS-SF), obtained from representative student survey
Change in decision-making (self-efficacy, future orientation) | Up to 36 months
  Score on the ZIMBARDO time perspective survey, Life Orientation Test - Revised (LOT-R), and other measures, obtained from representative student survey
Change in peer aggression | Up to 36 months
  Self-reported survey measures, obtained from representative student survey
Change in somatization | Up to 36 months
  Self-reported survey measures, obtained from representative student survey
Change in attention problems (hyperactivity) | Up to 36 months
  Self-reported survey measures, obtained from representative student survey
Change in interpersonal relationships | Up to 36 months
  Self-reported survey measures, obtained from representative student survey
Change in locus of control and anger management | Up to 36 months
  Self-reported survey measures, obtained from representative student survey
Change in empowerment | Up to 36 months
  Self-reported survey measures, obtained from representative student survey
Change in self-concept | Up to 36 months
  Self-reported survey measures, obtained from representative student survey
Change in social supports | Up to 36 months
  Self-reported survey measures, obtained from representative student survey
Change in perception of racial / cultural identity | Up to 36 months
  Self-reported survey measures, obtained from representative student survey

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No